CLINICAL TRIAL: NCT06515067
Title: Effect of Back Massage on ınfertılıty Stress, Sexual satısfactıon and marrıage Harmony ın ınfertılıty Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Emine Özge AVCI, PhD student, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 0000000
Record Dates: First submitted 2024-07-04; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Sexual Activity; Infertility; Stress
Keywords: infertility; back massage; sexual satisfaction
MeSH Terms: conditions — Sexual Behavior; Infertility; Orgasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): People in this group applied back massage
  Interventions: Other: back massage
- control group (Other): People in this group did not apply back massage
  Interventions: Other: no ıntervention

INTERVENTIONS:
Other: back massage — back massage
  Arms: study group
Other: no ıntervention — no ıntervention
  Arms: control group

SUMMARY:
This study aimed to investigate the effect of back massage on infertility stress, sexual satisfaction and marital harmony in infertile couples.

It aims to answer the question "Does back massage increase sexual satisfaction and marital harmony in infertile couples?" They will apply infertile chirt back massage and then answer survey questions about sexual satisfaction and marital harmony.

DETAILED DESCRIPTION:
Infertility is defined as the inability to become pregnant despite regular, unprotected sexual intercourse for 12 months. Infertility can cause decreased sexual satisfaction, deterioration of marital harmony and separation in couples. Massage with contact and touch can increase harmony between couples, reduce stress and contribute to increased sexual satisfaction. This study aimed to investigate the effect of back massage on infertility stress, sexual satisfaction and marital harmony in infertile couples.

The couples included in the study were divided into two groups: study and control groups. All patients completed the demographic information scale, The COMPI Coping Strategy Scales, Golombok Rust Sexual Satisfaction Scale and Marital Adjustment Scale. Back massage was taught to the couples in the study group and the spouses were allowed to perform back massage during the infertility treatment. No intervention was applied in the control group. A month later, the COMPI Coping Strategy Scales, Golombok Rust Sexual Satisfaction Scale and Marital Adjustment Scale were repeated on the fences. Mann Whitney u test, ki kare test and wilxon test used to analyze data.

Marital harmony and sexual satisfaction were found to be higher and stress levels were lower in couples who received back massage.

As a result, it has been shown that back massage has positive effects on infertility stress, sexual satisfaction and marital harmony in infertile couples.

ELIGIBILITY:
Inclusion Criteria:

Being 18 years or older, Being diagnosed with infertility, Being married and spouses living together, Being literate, There is no mental or psychological disorder/disability that would affect understanding and perception, Not having a problem that prevents massage (must not be an extremity amputee, should not have a fracture or dislocation, should not have an open wound)

Exclusion Criteria:

* Unable to communicate,
* Couples who do not want to participate in the research will not be included in the research.
* Those who have conditions that prevent massage (those with fever, wounds on their backs, individuals with tumors, the presence of an incomprehensible mass, those with orthopedic disorders, etc.) Exclusion Criteria for the Control Group
* Individuals who cannot be contacted and do not want to participate in the research will not be included in the research.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-11-26 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
İnfertility stress scale for measuring infertility stres | 2 mouths
  It is a scale developed by Schmidt (2006) to evaluate the stress experienced by infertile couples. The scale is a four-point Likert type (1: not at all, 4: very much), consists of 3 dimensions and 14 items.
Marital Adjustment Scale | 2 mounths
  The scale not only measures general marital satisfaction or quality, but also evaluates relationship style on issues such as expression of emotions, family budget, agreement or disagreement on issues such as sexuality and social rules, leisure activities, conflict resolution, and trust.
Golumbuok Rust Sexual Satisfaction Scale | 2 Mounths
  The scale is a measurement tool to evaluate the quality of sexual intercourse and sexual dysfunctions. The total score obtained gives a general idea about the quality of sexual functions, and the subscale scores provide more detailed information about the aspects of the relationship. There are two separate forms prepared for men and women, each consisting of 28 items.

SECONDARY OUTCOMES:
COMPI coping with infertility stress scale | 2 mouths
  The scale, developed to measure coping strategies with certain stressors related to infertility, consists of 19 items. In the scale, items 1 to 17 are evaluated on a 4-point Likert scale, and items 18 and 19 are evaluated on a 3-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: emine özge avcı, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes Üniversitei, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Background] Agarwal A, Baskaran S, Parekh N, Cho CL, Henkel R, Vij S, Arafa M, Panner Selvam MK, Shah R. Male infertility. Lancet. 2021 Jan 23;397(10271):319-333. doi: 10.1016/S0140-6736(20)32667-2. Epub 2020 Dec 10. PMID 33308486
- [Background] Alirezaei S, Ozgoli G, Alavi Majd H. Evaluation of Factors Associated with Sexual Function in Infertile Women. Int J Fertil Steril. 2018 Jul;12(2):125-129. doi: 10.22074/ijfs.2018.5193. Epub 2018 Mar 18. PMID 29707928
- [Background] Aourell M, Skoog M, Carleson J. Effects of Swedish massage on blood pressure. Complement Ther Clin Pract. 2005 Nov;11(4):242-6. doi: 10.1016/j.ctcp.2005.02.008. PMID 16290894

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT06515067/Prot_SAP_000.pdf